CLINICAL TRIAL: NCT06487507
Title: Metabolic Impact and Compliance of Controlled, Varying, Mediterranean Diets in Pre-Surgical Prostate Cancer Populations (PROVISIONS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Nima Sharifi, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20240052
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Fat Diet Group (Experimental): Participants in this group will receive a low fat Mediterranean diet for 2 weeks.
  Interventions: Behavioral: Low fat diet
- Lower Carbohydrate Mediterranean Diet Group (Experimental): Participants in this group will receive a lower carbohydrate Mediterranean diet for 2 weeks.
  Interventions: Behavioral: Lower carbohydrate diet

INTERVENTIONS:
Behavioral: Low fat diet — Prior to surgery, participants complete diet records for 7 days. After, participants will receive one shipment containing prepared meals (refrigerated, frozen and fresh) low fat Mediterranean that will be tested on this trial. The dietary intervention will be followed daily for two (2) weeks. Participants will complete a food frequency questionnaire to track food consumption. The diet will focus on including lean protein sources, high-quality fat and high-quality carbohydrate sources among others, and will limit refined sugars and high glycemic carbohydrates.
  Arms: Low Fat Diet Group
Behavioral: Lower carbohydrate diet — Prior to surgery, participants complete diet records for 7 days. After, participants will receive one shipment containing prepared meals (refrigerated, frozen and fresh) lower carbohydrate Mediterranean that will be tested on this trial. The dietary intervention will be followed daily for two (2) weeks. Participants will complete a food frequency questionnaire to track food consumption. The diet will focus on including lean protein sources, high-quality fat and high-quality carbohydrate sources among others, and will limit refined sugars and high glycemic carbohydrates.
  Arms: Lower Carbohydrate Mediterranean Diet Group

SUMMARY:
The study aims to investigate whether following a controlled Mediterranean-style diet prior to robotic-assisted radical prostatectomy surgery in patients diagnosed with prostate cancer affects fasting insulin levels and other values that can be measured in blood and tissue samples from surgery.

ELIGIBILITY:
Inclusion Criteria:

* Males 18 to 80 years old scheduled to undergo radical prostatectomy as per standard of care.
* BMI between 18.5 and 40
* Ability to read, write, speak, and understand English and/or Spanish.
* Ability to provide informed consent.
* Willingness to consume provided dietary interventions.
* Adequate organ and marrow function as assessed by treating clinician(s) which includes: White blood cell count (WBC) ≥2,500/microliter. Absolute neutrophil count (ANC) ≥1,500/microliter. Platelets ≥100,000/microliter. Hemoglobin ≥9 g/dL (transfusions permitted) Total bilirubin ≤1.5 x the institutional upper limit of normal (ULN). For subjects with Gilbert's disease ≤3.0 mg/dL. Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) ≤2.5 x institutional ULN. Creatinine clearance ≥51 ml/min as defined by Cockcroft-Gault equation.

Exclusion Criteria:

* Currently consuming a Mediterranean, lower carbohydrate, ketogenic, vegan, vegetarian, high fiber diet (14g fiber > per 1,000 Calories) and/or any supplements (including herbal), vitamins, minerals, that would interfere with diets being tested in the study as determined by dietitian and/or investigators as these diets are highly restrictive and may impact objectives/outcomes in the trial.
* Previous intolerability to fiber-rich diets.
* Colitis, Irritable Bowel Syndrome, or other gastrointestinal condition per clinician discretion.
* Food allergies or other major dietary restrictions.
* Receiving active medical treatment for Type I or Type II diabetes mellitus.
* Recent weight loss or gain (both intentional and unintentional) as defined by 5%+ body weight in the last 30 days.
* Undergone any type of weight loss surgery.
* Any medical contraindications as determined by investigators.
* History of diabetic ketoacidosis.
* History of Gout.
* Patients that are immunosuppressed (transplant history, on immunosuppression, etc.) as per clinician discretion.
* Gallbladder removed or plan to remove per clinician evaluation.
* Other malignancies actively receiving systemic treatment as per clinician evaluation.
* Previous treatment for prostate cancer.
* Previous history of pelvic radiation.
* Patients with impaired decision-making capacity.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients consuming Mediterranean diet | Up to 2 weeks
  Defined as the proportion of patients who consumed greater than 80% of provided calories using diet records.

SECONDARY OUTCOMES:
Change in fasting insulin | Baseline to 2 weeks
  Measured in milliliters
Change in high-sensitivity c-reactive protein | Baseline to 2 weeks
  Measured in milligrams per liter
Change in fasting glucose | Baseline to 2 weeks
  Measured in milligrams per deciliter
Change in blood pressure | Baseline to 2 weeks
  Measured in millimeters of mercury
Dietary behavior as measured by diet records questionnaire | Up to 2 weeks
  Measured in percentage of meals consumed by the participants
Number of treatment related adverse events | Up to 2 weeks
  Measured by fewer than three grade 3 adverse events using the NCI CTCAE version 6.0.

CONTACTS AND LOCATIONS:
Overall Officials: Nima Sharifi, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No